CLINICAL TRIAL: NCT01950273
Title: A Randomized, Double-blind, Parallel-arm, Phase I Study to Evaluate the Pharmacokinetics and Pharmacodynamics of BI 695500 vs. Rituximab (MabThera) Induction Immunotherapy as a First-line Treatment in Patients With Low Tumor Burden Follicular Lymphoma
Brief Title: Pharmacokinetics and Pharmacodynamics of BI 695500 vs. Rituximab as First Line-treatment in Patients With Low Tumor Burden Follicular Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1301.5; 2013-001904-12 (EudraCT Number)
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Results first posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab

ARMS (2):
- BI695500 (Experimental): BI695500, once a week for 4 weeks (4 administrations in total)
  Interventions: Drug: BI 695500
- MabThera (Active Comparator): MabThera, once a week for 4 weeks (4 administration in total)
  Interventions: Drug: MabThera

INTERVENTIONS:
Drug: BI 695500 — BI695500, once a week for 4 weeks (4 administrations in total)
  Arms: BI695500
Drug: MabThera — MabThera, once a week for 4 weeks (4 administrations in total)
  Arms: MabThera

SUMMARY:
The primary objective of the study is to assess the pharmacokinetic (PK) similarity of Boehringer Ingelheim (BI) 695500 vs. rituximab (MabThera®) in previously untreated patients with low tumor burden follicular lymphoma (LTBFL).

The secondary objective of the study is to evaluate the pharmacodynamics (PD), safety, and anti-tumor activity of BI 695500 vs. rituximab (MabThera®), as well as the presence of anti-drug antibodies (ADAs).

ELIGIBILITY:
Inclusion criteria:

* Must give written informed consent and be willing to follow this Clinical Trial Protocol.
* Male or female patients, at least 18 years of age at Screening.
* Histologically-confirmed, stage II - IV Non-Hodgkin's lymphoma (CD20+ FL of Grades 1, 2, or 3a).
* Low tumor burden according to the Groupe d'Etudes des Lymphomes Folliculaires (GELF) criteria - no nodal or extranodal involvement of more than 7 cm, no more than 3 nodal sites with a diameter >3 cm, no B symptoms (i.e., fever >38°C, weight loss - unexplained loss of >10 % body weight over the past 6 months, and sweats - the presence of drenching night sweats), no significant splenomegaly, no significant serious effusion, no complications such as organ compression, and less than 5x10^9/L circulating tumor cells.
* Availability of archived tumor sample prior to screening.
* Patients not previously treated for their FL.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Have at least 1 measurable lesion as per the International Working Group (IWG) criteria 2007 at Screening (lesion clearly measurable in at least 2 perpendicular dimensions; see Appendix 10.1 for further details).
* Adequate hematological function (unless abnormalities are related to lymphoma infiltration of the bone marrow) within 28 days prior to randomization, including:
* - hemoglobin =9.0 g/dL (=5.6 mmol/L).
* - absolute neutrophil count =1.5 × 10^9/L.
* - platelet count =100 × 10^9/L.
* Adequate renal and liver function:
* - serum creatinine <2.0 mg/dL (<176.8 micromol/L).
* - total bilirubin <2.0 mg/dL (<34 mcmol/L) except for patient with Gilbert's Syndrome or Hemolysis. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 x upper limit of normal (ULN) (<5 x ULN is acceptable if abnormalities are thought to be related to hepatic infiltration by FL).
* For participants of reproductive potential (males and females), use of a medically acceptable method of contraception during the trial, i.e., a combination of 2 forms of effective contraception (defined as hormonal contraception, intrauterine device, condom with spermicide, etc.). Females of childbearing potential (includes tubal ligation) and males with female partners of childbearing potential must also agree to use an acceptable method of contraception (see above) for 12 months following completion or discontinuation from the trial medication.

Exclusion criteria:

* Transformation to high-grade lymphoma (secondary to low-grade lymphoma).
* Presence or history of central nervous system lymphoma.
* Patients receiving current treatment with corticosteroids must not be receiving a dose exceeding 20 mg/day prednisone or equivalent.
* Patients with prior or concomitant malignancies within 5 years prior to screening except non-melanoma skin cancer, adequately treated carcinoma in situ of the cervix, adequately treated breast cancer in situ, localized prostate cancer stage T1c - provided that the patient underwent curative treatment, and remains relapse free.
* Major surgery (excluding lymph node biopsy) within 28 days prior to randomization.
* Active, chronic or persistent infection that might worsen with immunosuppressive treatment (e.g., Human Immunodeficiency Virus [HIV], Hepatitis C Virus [HCV], Herpes Zoster); positive for HIV or tuberculosis at Screening.
* Patients with serological evidence of Hepatitis B virus (HBV) infection. Patients seropositive because of HBV vaccine are eligible. HBV positive patients may participate following consultation with a hepatitis expert regarding monitoring and use of HBV antiviral therapy, and provided they agree to receive treatment as indicated.
* Serious underlying medical conditions, which, per the investigator's discretion, could impair the ability of the patient to participate in the trial (including but not limited to ongoing active infection, severe immunosuppression, uncontrolled diabetes mellitus, gastric ulcers, active autoimmune disease); patients who have significant cardiac disease, including but not limited to congestive heart failure of Class III or IV of the NYHA classification; uncontrolled angina or arrhythmia; any uncontrolled or severe cardiovascular or cerebrovascular disease.
* Known hypersensitivity or allergy to murine products.
* History of a severe allergic reaction or anaphylactic reaction to a biological agent or history of hypersensitivity to any component of the trial drug.
* Receipt of a live/attenuated vaccine within 12 weeks prior to the Screening Visit.
* Prior treatment with BI 695500 and/or rituximab.
* Patients who received any prior therapy using monoclonal antibodies will be excluded; this does not apply to other biological drugs such as growth factors or anticoagulants.
* Treatment within a clinical trial within 4 weeks prior to initiation of trial treatment. Patients who have received treatment with a drug that has not received regulatory approval for any indication within 4 weeks or a minimum of 5 half-lives, whichever is longer, of the initial dose of trial medication.
* Any other co-existing medical or psychological condition(s) that will preclude participation in the trial or compromise ability to give informed consent and/or comply with study procedures.
* Pregnancy or breast feeding. For women of childbearing potential, a positive serum pregnancy test at the Screening Visit.
* Patients who have significant cardiac disease, including but not limited to congestive heart failure of Class III or IV of the New York Heart Association (NYHA) classification; uncontrolled angina or arrhythmia; any uncontrolled or severe cardiovascular or cerebrovascular disease; or uncontrolled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-09-27 (Actual); Primary Completion 2015-12-22 (Actual); Study Completion 2015-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (29):
- The Canberra Hospital, Canberra, Migration Data, Australia
- AKH - Medical University of Vienna, Vienna, Austria
- Belgium (3):
  - Brussels - UNIV St-Luc, Brussels
  - UZ Leuven, Leuven
  - Namur - HOSP Ste-Elisabeth, Namur
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Czechia (3):
  - University Hospital Brno, Brno
  - University Hospital Ostrava, Ostrava-Poruba
  - Vseobecna fakultni nemocnice V Praze, Prague
- France (5):
  - INS Bergonié, Bordeaux
  - HOP Morvan, Brest
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - HOP Haut-Lévêque, Pessac
  - Hôpital la Milétrie - CHU Poitiers, Poitiers
- Germany (5):
  - Gesundheitszentrum Wetterau gGmbH, Bad Nauheim
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Haemato-Onkologie Hamburg, Hamburg
  - Klinikum Kassel GmbH, Kassel
- General Hospital of Athens "G. Gennimatas", Athens, Greece
- Semmelweis University, 1st Dept. Internal Medicine, Budapest, Hungary
- Auckland Clinical Studies Ltd, Auckland, New Zealand
- Oncol Centre M Sklodowska-Curie, Dept of Lung & Chest Cancer, Warsaw, Poland
- Russia (2):
  - BHI of Omsk region - Clinical Oncology Dispensary, Omsk
  - St. Petersburg GUZ City Clinical Oncology Dispensary, Saint Petersburg
- Spain (4):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Puerta del Mar, Cadiz
  - Fundación Jiménez Díaz, Madrid
  - Hospital Virgen del Rocío, Seville

RESULTS

PARTICIPANT FLOW:
Groups:
- BI 695500: The subjects received BI 695500 (Test)/100 mg/10 mL concentrate for solution for infusion at 375 mg/m2 once a week for 4 weeks (for a total of 4 dosages administered on Days 1, 8, 15, and 22) by intravenous (IV) infusion.
- Rituximab (MabThera®): The subjects received Rituximab (MabThera® (Reference))/100 mg/10 mL and 500 mg/50 mL concentrate for solution for infusion at 375 mg/m2 once a week for 4 weeks (for a total of 4 dosages administered on Days 1, 8, 15, and 22) by IV infusion.
Period: Overall Study
Arm/Group | BI 695500 | Rituximab (MabThera®)
Started | 49 | 46
Completed | 45 | 46
Not Completed | 4 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other not defined above | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS): The patients who received at least one dose of trial medication and classified as per treatment received.
Groups:
- BI 695500: The subjects received BI 695500/100 mg/10 mL concentrate for solution for infusion at 375 mg/m2 once a week for 4 weeks (for a total of 4 dosages administered on Days 1, 8, 15, and 22) by intravenous (IV) infusion.
- Rituximab (MabThera®): The subjects received Rituximab (MabThera®)/100 mg/10 mL and 500 mg/50 mL concentrate for solution for infusion at 375 mg/m2 once a week for 4 weeks (for a total of 4 dosages administered on Days 1, 8, 15, and 22) by IV infusion.
- Total: Total of all reporting groups
Arm/Group | BI 695500 | Rituximab (MabThera®) | Total
Number analyzed (Participants) | 49 | 46 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (12.44) | 58.4 (11.48) | 59.0 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 26 | 19 | 45

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration (AUC) Time Curve of BI 695500 and Rituximab (MabThera®) Over the First Dosing Interval (Pre-infusion on Day 1 to Pre-infusion on Day 8)
Description: This outcome measure presents area under the concentration time curve of BI 695500 and Rituximab (MabThera®) over the first dosing interval (pre-infusion on Day 1 to pre-infusion on Day 8) (AUCDay 1-Day 8) for assessment of PK (Pharmacokinetics) similarity.
Time Frame: Blood samplings were done at pre-infusion and at end of infusion at 1, 2, and 4 hours from end of infusion 1, and at 24, 48, 72, 96 and 168 hours from start of infusion 1.
Population: The PK analysis Set Inferential (PKSI) used for inferential analysis of PK parameters, consisted of all randomized subjects who received at least one dose of trial medication and had an estimable primary PK parameter value and were without important protocol deviations that would significantly affect the PK of BI 695500 or Rituximab (MabThera®).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/millilitre (µg*h/mL)
Arm/Group | BI 695500 | Rituximab (MabThera®)
Number analyzed (Participants) | 46 | 43
microgram*hour/millilitre (µg*h/mL) | 15700 (69.8) | 17600 (27.9)
Statistical Analysis 1: Comparison: BI 695500 vs Rituximab (MabThera®); Test type: Non-Inferiority or Equivalence — Standard equivalence limit 80% to 125%; Least Squares (LS) mean ratio = 89.53, 90% CI 2-sided [75.42 to 106.29] — Ratio of the adjusted geometric means calculated as (LS mean ratio of BI 695500/Rituximab (MabThera®))

2. Secondary Outcome: AUC of BI 695500 and Rituximab (MabThera®) Over the Fourth Dosing Interval (Pre-infusion on Day 22 to Day 29) (AUC Day 22-Day 29)
Description: This outcome measure presents area under the concentration of BI 695500 and Rituximab (MabThera®) over the fourth dosing interval (pre-infusion on Day 22 to Day 29).
Time Frame: Blood samplings were done at pre-infusion and at end of infusion at 1, 2, and 4 hours from end of infusion 4, and at 24, 48, 72, 96 and 168 hours from start of infusion 4.
Population: The PK analysis Set Inferential (PKSI) used for inferential analysis of PK parameters, consisted of all randomized subjects who received at least one dose of trial medication and had estimable primary PK parameter value and were without important protocol deviations that would significantly affect the PK of BI 695500 or Rituximab (MabThera®).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/millilitre (µg*h/mL)
Arm/Group | BI 695500 | Rituximab (MabThera®)
Number analyzed (Participants) | 40 | 43
microgram*hour/millilitre (µg*h/mL) | 41700 (32.3) | 44300 (24.8)
Statistical Analysis 1: Comparison: BI 695500 vs Rituximab (MabThera®); Test type: Non-Inferiority or Equivalence — Standard equivalence limit 80% to 125%; Least Squares (LS) means ratio = 94.60, 90% CI [85.04 to 105.23] — Ratio of the adjusted geometric means calculated as (LS mean ratio of BI 695500/Rituximab (MabThera®))

3. Secondary Outcome: Maximum Measured Concentration of BI 695500 and Rituximab (MabThera®) in Plasma (Cmax) Following Dose 1
Description: This outcome measure presents maximum measured concentration of BI 695500 and Rituximab (MabThera®) in plasma (Cmax) following Dose 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/millilitre (µg/mL)
Arm/Group | BI 695500 | Rituximab (MabThera®)
Number analyzed (Participants) | 46 | 44
microgram/millilitre (µg/mL) | 207.882 (58.5) | 228.802 (25.0)
Statistical Analysis 1: Comparison: BI 695500 vs Rituximab (MabThera®); Test type: Non-Inferiority or Equivalence — Standard equivalence limit 80% to 125%; Least Squares (LS) means ratio = 89.94, 90% CI 2-sided [77.62 to 104.23] — Ratio of the adjusted geometric means calculated as (LS mean ratio of BI 695500/Rituximab (MabThera®))

4. Secondary Outcome: Maximum Measured Concentration of Rituximab (MabThera®) and BI 695500 in Plasma (Cmax) Following Dose 4
Description: This outcome measure presents maximum measured concentration of Rituximab (MabThera®) and BI 695500 in plasma (Cmax) following Dose 4.
Time Frame: Blood samplings were done at pre-infusion and at end of infusion at 1, 2, and 4 hours from end of infusion 4, and at 24, 48, 72, 96, 168, 336, 672, 1344, 2016 and 2880 hours from start of infusion 4.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/millilitre (µg/mL)
Arm/Group | BI 695500 | Rituximab (MabThera®)
Number analyzed (Participants) | 39 | 42
microgram/millilitre (µg/mL) | 397.080 (23.1) | 412.190 (18.1)
Statistical Analysis 1: Comparison: BI 695500 vs Rituximab (MabThera®); Test type: Non-Inferiority or Equivalence — Standard equivalence limit 80% to 125%; Least Squares (LS) means ratio = 97.65, 90% CI 2-sided [90.45 to 105.42] — Ratio of the adjusted geometric means calculated as (LS mean ratio of BI 695500/Rituximab (MabThera®))

5. Secondary Outcome: Area Under the Depletion-time Curve of the Cluster of Differentiation (CD)19+ B-cell Count (% Change From Baseline (CFB)) in Peripheral Blood From Pre-infusion on Day 1 Until Last Measurement on Day 8 (Pre-infusion)
Description: This outcome measure presents area under the depletion-time curve of the CD19+ B-cell count (% change from baseline) in peripheral blood from pre-infusion on Day 1 until last measurement on Day 8 (pre-infusion) (AUC Day 1-Day 8, CD19+).
Time Frame: Blood samplings were done at pre-infusion and at end of infusion at 1, 2, and 4 hours from end of infusion, and at 24, 48, 72, 96 and 168 hours from start of infusion.
Population: The PK analysis Set Descriptive (PKSD) consisted of all randomized subjects who received at least one dose of trial medication BI 695500 or Rituximab [MabThera®], had at least one post-treatment PK concentration value and were without important protocol deviations that would significantly affect the PK of BI 695500 or Rituximab (MabThera®).
Measure: Mean (Standard Deviation); unit: Percentage CFB of CD19+ B-cells*hour
Arm/Group | BI 695500 | Rituximab (MabThera®)
Number analyzed (Participants) | 32 | 41
Percentage CFB of CD19+ B-cells*hour | -16895.2 (1016.9) | -17064.4 (1403.2)
Statistical Analysis 1: Comparison: BI 695500 vs Rituximab (MabThera®); Test type: Superiority or Other; Mean Difference (Final Values) = 249.2, 90% CI 2-sided [-210.6 to 709] — Mean difference calculated as BI 695500-Rituximab (MabThera®)

6. Secondary Outcome: Change From Baseline (%) of CD19+ B-cells in Peripheral Blood Measured After Seven Days on Day 8 (Day 8 Pre-infusion Time Point)
Description: This outcome measure presents percent change from baseline of CD19+ B-cells in peripheral blood, measured after 7 days (i.e., Day 8 pre-infusion time point) (PCFBpre,2 CD19+).
Time Frame: Blood sampling was done at 168 hours from start of infusion.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage (%) CFB of CD19+ B-cells
Arm/Group | BI 695500 | Rituximab (MabThera®)
Number analyzed (Participants) | 33 | 42
Percentage (%) CFB of CD19+ B-cells | -99.2 (1.7) | -98.8 (4.2)

7. Secondary Outcome: Overall Response Rate (ORR) (Complete Response (CR) Plus Partial Response (PR)) Evaluated Approximately One Month After Last Dose of BI 695500 or Rituximab (MabThera®)
Description: Overall Response Rate (ORR) comprised Complete Response (CR) plus Partial Response (PR) evaluated approximately one month after last dose of BI 695500 or Rituximab [MabThera®]. Overall Response as defined by the revised International Working Group (IWG) Criteria 2007, using the Investigator's assessment.
Time Frame: at Day 50.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of subjects
Arm/Group | BI 695500 | Rituximab (MabThera®)
Number analyzed (Participants) | 22 | 25
Percentage of subjects | 44.9 | 54.3
Statistical Analysis 1: Comparison: BI 695500 vs Rituximab (MabThera®); Test type: Superiority or Other; Mean Difference (Final Values) = -9.4, 95% CI 2-sided [-29.4 to 11.1] — Difference in ORR calculated as ORR (BI695500) - ORR (MabThera®). The confidence interval represented is 95% difference in proportions

8. Secondary Outcome: Percentage of Patients With Treatment Emergent Adverse Events (TEAEs) Selected for Comparability Assessment of BI 695500 and Rituximab (MabThera®)
Description: This outcome measure presents percentage of patients with Treatment Emergent Adverse Events (TEAEs) selected for comparability assessment of BI 695500 and Rituximab (MabThera®).
Time Frame: Adverse Events (AEs) that started or worsened on or after the first dose of study medication and prior to the last date of study medication + 4 months (120 days) inclusive.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients
Arm/Group | BI 695500 | Rituximab (MabThera®)
Number analyzed (Participants) | 18 | 16
Percentage of patients | 36.7 | 34.8
Statistical Analysis 1: Comparison: BI 695500 vs Rituximab (MabThera®); Test type: Superiority or Other; Median Difference (Final Values) = 2.0, 95% CI 2-sided [-18.0 to 22.1] — Difference in TEAE incidence calculated as BI695500 - TEAE incidence (MabThera®). The confidence interval represented is 95% difference in proportions

ADVERSE EVENTS:
Time Frame: From first drug administration until 142 days after last drug administration, up to 156 days.
Arm/Group | BI 695500 | Rituximab (MabThera®)
Serious Adverse Events (participants affected / at risk) | 4/49 | 3/46
Other Adverse Events (participants affected / at risk) | 25/49 | 28/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695500 (N=49) | Rituximab (MabThera®) (N=46)
Vertigo (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Anaphylactoid reaction (Immune system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abortion induced (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695500 (N=49) | Rituximab (MabThera®) (N=46)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 7
Asthenia (General disorders) | 6 | 1
Fatigue (General disorders) | 2 | 4
Pyrexia (General disorders) | 4 | 5
Alanine aminotransferase increased (Investigations) | 5 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 3
Blood cholesterol increased (Investigations) | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 3 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Headache (Nervous system disorders) | 5 | 7
Insomnia (Psychiatric disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 7
Hypertension (Vascular disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes